CLINICAL TRIAL: NCT06072625
Title: The Effect of Enteral Organic Extra Virgin Olive Oil Supplementation in Premature Babies on Postnatal Growth and Premature Morbidities
Brief Title: Enteral Feeding of Premature Babies and Olive Oil Supplementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Bayram Ali DORUM, Head of Division of Neonatology, Associate Professor, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BCH-2023-12/8
Record Dates: First submitted 2023-09-13; First posted 2023-10-10 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Premature; Olive Oil; Enteral Feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive oil group (Active Comparator): Babies who have fully enteral feeding will take oral, 1 ml/kg/day of extra virgin olive-oil
  Interventions: Dietary Supplement: Extra virgin organic olive oil (ULTRA PREMIUM)
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Extra virgin organic olive oil (ULTRA PREMIUM) — Babies who have fully enteral feeding will take oral, 1 ml/kg/day of extra virgin olive-oil
  Arms: Olive oil group

SUMMARY:
It is a two-arm prospective interventional study. 40 babies in both groups will be enrolment in the study. In the intervention group, babies will take 1 ml/kg/day of the study product (ULTRA PREMIUM) after full enteral feeding.

Supplementation will continue until discharge or the 36th week. Blood samples will be taken for serum Total antioxidant capacity and Malondialdehyde levels before the intervention and on the 14th day of the control group. At the end of the study, serum will be taken again for control values.

Daily lipid intake amounts will be recorded through breast milk analysis. Lipid profile will be monitored weekly The growth parameters of babies will be monitored daily It will be evaluated at the end of the study in terms of ROP, BPD, and NEC. At the end of the study, the data of babies in both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies born at 32 weeks or less
* Babies who tolerate full enteral feeding at the before end of the second week
* Babies given consent by their parents -

Exclusion Criteria:

* Having a congenital or genetic anomaly

Ages: 14 Days to 40 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who completed the study | 15 months
  To enrolment of 40 babies in the study in both groups
Postnatal growth retardation rates | 18 months
  Daily weight intake amounts of babies in both groups

SECONDARY OUTCOMES:
Frequency and severity of retinopathy of prematurity | 18 months
  Frequency and severity of retinopathy of prematurity

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No